CLINICAL TRIAL: NCT07053852
Title: Activation of Ameluz With BBL HEROic for the Treatment of Actinic Keratoses and Photodamage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sherrif Ibrahim (Other)
Collaborators: Sciton (Industry); Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor-Investigator, Sherrif Ibrahim, Principal Investigator, Rochester Dermatologic Surgery
Organization: Rochester Dermatologic Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF-BBL-01
Record Dates: First submitted 2025-02-05; First posted 2025-07-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Actinic Keratoses; Photodamage
Keywords: aging face; actinic keratosis; BBL; PDT; photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Two PDT treatments (Experimental): Each subject will receive 2 treatments of photodynamic therapy using Ameluz and HEROic BBL to treat facial AK and signs of photodamage.
  Interventions: Drug: Ameluz; Device: Sciton HEROic

INTERVENTIONS:
Drug: Ameluz — broad band light (BBL) with the use of Ameluz
Device: Sciton HEROic — Each subject will receive 2 treatments of photodynamic therapy using Ameluz and HEROic BBL to treat facial AK and signs of photodamage.
  Other Names: BBL

SUMMARY:
To provide a treatment of both actinic keratoses and photodamage within one treatment.

DETAILED DESCRIPTION:
To demonstrate that treatment of actinic keratoses and photodamage with a combination of Ameluz and Broad Band Light (BBL) will lead to an improvement in facial precancerous change and signs of photodamage.

ELIGIBILITY:
Inclusion Criteria:

* Over 18yrs of age
* Willingness to participate in all required study activities and visits
* Willingness to sign the informed consent form
* Visible and palpable signs of diffuse actinic damage and actinic keratoses of mild to moderate severity located on the face
* Significant signs of photoaging, evaluated by investigator, that include any or all the following:

  * Dyspigmentation
  * Solar lentigines
  * Telangiectasias
  * Diffuse erythema
  * Roughness and other textural changes
  * Fine lines
  * Wrinkles
  * Actinic bronzing

Exclusion Criteria:

* Subject who is unable and unwilling to provide consent for study schedule and procedures
* Subject who is pregnant or trying to become pregnant during the study
* Subjects using any topical treatment on their AKs; must stop at least one month prior
* Subjects currently undergoing cancer treatment with medical or radiation therapy
* Subjects with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material
* Subjects with history of a photosensitivity disease, such as porphyria cutanea tarda

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Percentage of clearance of actinic keratoses | 2 months
  Percentage of actinic keratosis lesion clearance at 1 and 2 months after 2 treatments with the combination of Ameluz and BBL on the face.
Cosmetic outcomes | 2 months
  Cosmetic outcomes in photoaging of the face evaluated by Subject and Investigator Global Aesthetic Improvement Scale (GAIS) at 1 and 2 months post last PDT.
  Scale: Very Satisfied (better than expected), Satisfied (as expected), Unsatisfied (worse than expected)

SECONDARY OUTCOMES:
Percentage of clearance of actinic keratoses | 2 months
  Percentage of actinic keratosis lesion clearance at 1 and 2 months after 2 treatments with the combination of Ameluz and BBL on the face using a Visia camera analysis.
Cosmetic outcomes | 2 months
  Cosmetic outcomes in photoaging of the face evaluated a Visia camera analysis at 1 and 2 months post last PDT

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Dermatologic Surgery, Victor, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided